CLINICAL TRIAL: NCT05519826
Title: A Retrospective, Observational Study to Collect Clinical Safety and Performance Data of POLYMAILLE® EXTRA THIN Vascular Prothesis
Status: Completed | Type: Observational
Sponsor: Perouse Medical (Industry)
Collaborators: Eclevar Medtech (Industry)
Responsible Party: Sponsor
Other Study IDs: PMET-2022-01
Record Dates: First submitted 2022-08-26; First posted 2022-08-29 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Aneurysm Abdominal; Peripheral Aneurysms; Arterial Disease Occlusive; Prothesis
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Arterial Occlusive Diseases | interventions — Vascular Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Vascular surgery — POLYMAILLE® EXTRA THIN vascular prostheses are indicated for replacement or bypass of arteries presenting aneurysm or obliterative arterial disease. Their indication is restricted to abdominal and peripheral surgery not crossing the knee flexion crease.
  Abdominal vascular surgery includes aorto-iliac and/or aorto-femoral vascular repair, i.e. graft implantation with proximal anastomosis to abdominal aorta (supra and/or infra-renal).
  Peripheral vascular surgery includes peripheral arteries repair, i.e. graft implantation with no aortic anastomosis, and/or extra-anatomic vascular repair such as axillo-femoral and/or crossover bypass (femoro-femoral and/or ilio-femoral) and/or femoro-popliteal bypass above the knee.

SUMMARY:
The purpose of this PMCF study is to evaluate a minimum of 125 subjects in 1 or 2 sites in France at least 1-year follow-up after surgery until a maximum of 5 years in the indication of abdominal and peripheral arterial surgery not crossing the knee flexion crease.

the objectives of the evaluation will describe safety and performance of POLYMAILLE® EXTRA THIN.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all the following inclusion criteria in order to be eligible for inclusion in the study:

Patient has a minimum of 1-year post-operative follow-up data available, or complete data to death

Exclusion Criteria:

* Patients who refused the collection of their personal data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient population conditions that may indicate abdominal and/or peripheral vascular open surgical repair with implantation of a POLYMAILLE EXTRA THIN vascular graft include:
  * Peripheral arterial diseases (PAD), characterized by reduced blood flow to the lower extremities, which may be categorized as:
    * Intermittent claudication (IC)
    * Chronic limb-threatening ischemia (CLTI)
    * Acute limb ischemia (ALI)
  * Peripheral arterial aneurysms, characterized by a permanent localized (i.e., focal) modification of the parallelism of the vessel walls, which may be categorized by the following location:
    * Iliac arterial aneurysms (IAA)
    * Femoral arterial aneurysms (FAA)
    * Popliteal arterial aneurysms (PAA)
Sampling Method: Probability Sample
Enrollment: 373 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Primary performance endpoint | 1 year
  primary patency rate
Primary safety endpoint | 1 year
  limb salvage rate

SECONDARY OUTCOMES:
Procedural success rate | 5 years
  * Ability to use with no need for replacement by another device and,
  * Effective vascular flow restoration after procedure and,
  * In case of aneurysm, exclusion of aneurysmal portion after procedure.
Primary patency rate | 5 years
  patent grafts without any procedure or intervention of the conduit itself
Primary assisted patency rate | 5 years
  rate of patent grafts, with or without procedure or intervention of the conduit itself after device implantation, such as endovascular balloon angioplasty or anastomotic revision, however with graft never thrombosed (graft occlusion)
-Secondary patency rate | 5 years
  rate of patent grafts, with or without procedure or intervention of the conduit itself after device implantation, such as endovascular balloon angioplasty or anastomotic revision, lysis and/or thrombectomy
Device Failure | 5 years
  * Uncontrolled blood leakage from device
  * Loss of structural integrity, e.g. rupture and/or exaggerated dilation (> 50 %)
  * Occlusion of the device
  * Total or partial replacement of the device required
Mortality rate | 5 years
  freedom % from death
Limb salvage rate | 5 years
  freedom % from target limb major amputation
Adverse events | 5 years
  any documented adverse events, including anticipated (as listed in section 6.2) and non-anticipated adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No